CLINICAL TRIAL: NCT03402308
Title: Effect of Schisandra Chinensis Extract on Musculoskeletal Biomakers in Relatively Sarcopenic Adults: a Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Effect of Schisandra Chinensis Extract on Musculoskeletal Biomakers in Relatively Sarcopenic Adults: a RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Integrated Research Institute for Natural Ingredients and Functional Foods (IRINIF), Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2017-010
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Muscular Sarcoidosis
MeSH Terms: interventions — schizandrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schisandra chinensis extract group (Experimental): This group takes Schisandra chinensis extract for 12 weeks
  Interventions: Dietary Supplement: Schisandra chinensis extract
- Placebo group (Placebo Comparator): This group takes placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Schisandra chinensis extract — Schisandra chinensis extract 1,000 mg/day for 12 weeks
  Arms: Schisandra chinensis extract group
Dietary Supplement: Placebo — Starch placebo 1,000 mg/day for 12 weeks
  Arms: Placebo group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of the SCE on muscle strength, muscle mass, and muscle function in healthy adults for 12 weeks.

DETAILED DESCRIPTION:
Previous studies have indicated that Schisandra chinensis extract (SCE) may have the ability to prevent skeletal muscle atrophy. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of the SCE on muscle strength, muscle mass, and muscle function in healthy adults; the safety of the compound are also evaluate. The Investigators examine the peak torque/body weight at 60°/s knee extension, handgrip strength, skeletal muscle mass, physical performance, and metabolic parameters at baseline, as well as after 4 and 12 weeks of intervention. Fifty-four healthy adults were administered either 1,000 mg of SCE or a placebo each day for 12 weeks;

ELIGIBILITY:
Inclusion Criteria:

* <110% of the standard lean body mass as measured using the body composition analyzer InBody 720)
* Body-mass index (BMI) ranging from 18.5 to 30.0 kg/m2

Exclusion Criteria:

* Abnormal liver or renal function (i.e., serum aminotransferase activity > 60 IU/L and serum creatinine concentrations > 1.2 mg/dL)
* Diabetes (diagnosed clinically or fasting glucose level > 126 mg/dL)
* History of fracture during the previous year
* Uncontrolled hypertension
* History of serious cardiac disease such as angina or myocardial infarction
* History of gastrectomy
* History of medication for psychiatric disease
* Administration of oriental medicine including herbs within the past 4 weeks
* Evidence of relatively high skeletal mass (more than 110% of the standard lean body mass as measured using the body composition analyzer InBody 720)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
muscle strength | 12 weeks
  the peak torque/body weight at 60°/s knee extension

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Pusan, Ami-dong, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cho YH, Lee SY, Lee CH, Park JH, So YS. Effect of Schisandra chinensis Baillon extracts and regular low-intensity exercise on muscle strength and mass in older adults: a randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2021 Jun 1;113(6):1440-1446. doi: 10.1093/ajcn/nqaa447. PMID 33710261